CLINICAL TRIAL: NCT01867749
Title: Group Interpersonal Psychotherapy for Treatment of Major Depressive Disorder Following Perinatal Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Dr. Jennifer Johnson, Associate Professor (Research), Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5R34MH086682-03 (NIH); 5R34MH086682-03 (NIH)
Record Dates: First submitted 2013-05-28; First posted 2013-06-04 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Major Depressive Disorder; Miscarriage; Stillbirth; Neonatal Death
Keywords: Major Depressive Disorder (MDD); Miscarriage; Stillbirth; Neonatal death; Interpersonal psychotherapy; Group Therapy; Coping with Depression (CWD)
MeSH Terms: conditions — Depressive Disorder, Major; Abortion, Spontaneous; Stillbirth; Perinatal Death | interventions — Coping Skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Interpersonal Psychotherapy (IPT-G) (Experimental): Participants in the IPT-G condition will receive 12 group therapy sessions over 2 weeks as well as 2 individual (pre-group and 1-month booster sessions). In addition, 3 of the 12 group sessions will invite women to include their partners or other support people to bolster the woman's social support system and to reduce conflicts over how to react to the loss. This study adapted IPT for treatment of depression after perinatal loss.
  Interventions: Behavioral: Group Interpersonal Psychotherapy (IPT-G)
- Coping with Depression (CWD) (Active Comparator): The Coping with Depression (CWD) course is a highly structured, manualized psycho-educational group treatment for MDD. The course content is cognitive-behavioral in nature and is designed to train skills that can be used in the alleviation of depression. The skill modules focus on relaxation, cognitive skills, and behavioral activation. CWD will consist of an individual pre-group interview, 12 group therapy sessions over 12 weeks and a 1-month individual booster session to provide an identical treatment dose as the experimental condition.
  Interventions: Behavioral: Coping with Depression (CWD)

INTERVENTIONS:
Behavioral: Group Interpersonal Psychotherapy (IPT-G)
  Other Names: IPT-G
  Arms: Group Interpersonal Psychotherapy (IPT-G)
Behavioral: Coping with Depression (CWD)
  Other Names: CWD
  Arms: Coping with Depression (CWD)

SUMMARY:
The purpose of this study is to conduct a randomized pilot trial in a sample of 60 women who meet criteria for Major Depressive Disorder (MDD) 1-18 months after a perinatal loss to demonstrate the feasibility of the proposed recruitment methods and research design, of the therapist training methods, and of delivering the adapted Interpersonal Psychotherapy group treatment.

The investigators would like to examine preliminary evidence for the following hypotheses:

* Perinatal-loss specific IPT-G will be more acceptable to women who experience MDD following perinatal loss than will Coping with Depression (CWD).
* Perinatal-loss specific IPT-G will result in reduced time to remission from MDD and reduced depressive symptoms relative to CWD.
* Perinatal-loss specific IPT-G will result in increased social support and social functioning, reduced couple distress, and reduced grief relative to CWD.

ELIGIBILITY:
Inclusion Criteria:

* Current Major Depressive episode.
* Experience perinatal loss 1-18 months prior to intake (including early and late fetal death and the death of a live born neonate within the first 28 days).

Exclusion Criteria:

* Untreated thyroid difficulties (TSH levels out of the normal range).
* Anemia (hemoglobin or hematocrit out of the normal range).
* Onset of current major depressive episode prior to news of difficulties with the pregnancy or health risk to the infant (women with prior episodes will be included).
* Current or past diagnosis of bipolar I disorder, schizophrenia or other psychotic disorder.
* Primary diagnosis of substance dependence or eating disorder.
* Acute suicidal or homicidal risk.
* Non-stable course of antidepressant medication or psychotherapy (i.e., beginning or changing dose of either within the previous 8 weeks).
* Any IPT or cognitive-behavioral treatment in the previous 8 weeks.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2010-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Treatment Acceptability | Post Treatment (12 Weeks)
  Treatment acceptability measured by the End of Treatment Questionnaire and the client satisfaction questionnaire.
Reduced time to remission from major depressive disorder (exploratory in this underpowered feasibility/acceptability study) | Survival analysis
  We will calculate the effect size and confidence intervals for time to remission from depressive episode. Remission will be defined as number of weeks until Hamilton Rating Scale for Depression score of 7 or less. Recovery from major depression is an exploratory aim; it will be defined as 8+ consecutive weeks on the Longitudinal Interval Follow-up Evaluation PSR scores of 1 or 2. Exploratory tests for differences between conditions will use Cox regression, with initial HRSD scores as a covariate.
Reduction in depressive symptoms (exploratory in this underpowered feasibility/acceptability study) | Slopes over time
  We will calculate the effect sizes and confidence intervals for reduction in depressive symptoms using HRSD and BDI-II scores. Exploratory tests for differences between conditions will use HLM with baseline scores as covariates.

SECONDARY OUTCOMES:
Perceived Social Support | Slope over time: Baseline, 4 Weeks, 8 Weeks, 12 Weeks, 3 Months, 6 Months
  We will calculate effect sizes and confidence intervals for improvement in social support and social functioning using the Multidimensional Scale of Perceived Social Support and the Social Adjustment Scale. Exploratory tests for differences between conditions will use HLM with baseline scores as covariates.
Couple Distress | Slope over time: Baseline, 4 Weeks, 8 Weeks, 12 Weeks, 3 Months, 6 Months
  Social adjustment as measured by the Dyadic Adjustment Scale (DAS). We will calculate effect sizes and confidence intervals for reduction in couple distress using the DAS. Exploratory tests for differences between conditions will use HLM with baseline DAS scores as a covariate.
Grief | Slope over time: Baseline, 4 Weeks, 8 Weeks, 12 Weeks, 3 Months, 6 Months
  Grief as measured by the Perinatal Bereavement Grief Scale and the Inventory of Complicated Grief. We will calculate effect sizes and confidence intervals for reduction in grief using the PBGS and ICG. Exploratory tests for differences between conditions will use HLM with baseline scores as covariates. Although not the primary focus of this study, we will also calculate the NNT for prevention of complicated grief diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E. Johnson, Ph.D., Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States